CLINICAL TRIAL: NCT00922558
Title: Evaluation of Postural Control in Children Using Tetra Axial Posturography
Acronym: tetrax1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Dan Nemet M.D.,, Meir Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MeirMc068-09CTIL
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2009-06

CONDITIONS: Normal Children
Keywords: tetra-axiametric posturography; postural control; tetrax; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal children (No Intervention): Normal children ages 5-12 years.
  Interventions: Other: Evaluation of postural control
- postural control (Experimental)
  Interventions: Other: Evaluation of postural control

INTERVENTIONS:
Other: Evaluation of postural control — Children will be measured once using a Tetra-aximetric posturography method

SUMMARY:
Tetra-ataxiametric posturography is based on the measurement and computerized elaboration of electronic signals emitted by four footplates, one for each heel and toe, respectively. These are sensitive to vertical pressure produced by a subject standing straight but in various positions (feet parallel, in tandem, eyes closed, on pads, etc.). The method yields additional parameters not obtained by the traditional monoplate stabilometers, namely, weight-distribution patterns and correlation among six combinations of paired outputs from the two heels, two toes, heel/toe of each foot, and the two diagonals (tetra-ataxiametric synchronizations). Comparing age-matched learning disabled, mentally retarded, autistic, and hearing impaired (with and without labyrinthine hypofunction) with normal children, significant and clinically meaningful differences were detected between the Tetra-ataxiametric measures of stability, interaction between Fourier Spectral Power Ranges of body sway, weight distributions, and synchronizations of toe parts. The same parameters correlated significantly with cognitive school readiness in normal populations. While the stability and spectral quotients show significant developmental changes, weight distribution and toe synchronisations are stable from 5 years onwards. The method is suitable for young subjects and attractive to children who may ordinarily be reluctant to cooperate, such as the autistic ones. The equipment is portable and tests can be conveniently carried out in a child's familiar educational setting.

DETAILED DESCRIPTION:
Recently a new pediatric software was introduced for the TETRAX device. The goal of the present study is to create normative data for children starting at preschool age using the newly developed software. Four hundred and 80 children between the ages of 5 and 12 years old will be examined following informed consent from the children and their legal guardian.

ELIGIBILITY:
Inclusion Criteria:

* age 5-12 years
* healthy

Exclusion Criteria:

* children with known disturbances in bone, muscle of nervous systems
* children using medications that may cause problems in balance or coordination

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Creation of normal baseline data | one year

SECONDARY OUTCOMES:
evaluation of a new analysis software | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Pediatrics, Meir Medical Center, Sackler School of Medicine, Tel Aviv University
Locations (1):
- Reoven Cohen-Raz, Jerusalem, Israel